CLINICAL TRIAL: NCT01455857
Title: Phase 3, Randomized, Double-Blind, Placebo-Controlled, Multi-Center Study to Evaluate the Efficacy, Safety and Tolerability of ITCA 650 in Patients With Type 2 Diabetes
Brief Title: A Study to Evaluate ITCA 650 for the Treatment of Type 2 Diabetes
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Intarcia Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ITCA 650-CLP-103
Record Dates: First submitted 2011-10-18; First posted 2011-10-20 (Estimated); Last update posted 2015-08-18 (Estimated); Status verified 2015-07

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Exenatide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- ITCA 650 40 mcg/day (Experimental)
  Interventions: Drug: ITCA 650
- ITCA 650 60 mcg/day (Experimental)
  Interventions: Drug: ITCA 650
- ITCA placebo (Placebo Comparator)
  Interventions: Other: ITCA placebo

INTERVENTIONS:
Drug: ITCA 650 — ITCA 650 is exenatide in DUROS
  Arms: ITCA 650 40 mcg/day; ITCA 650 60 mcg/day
Other: ITCA placebo — Formulation in DUROS (no exenatide)
  Arms: ITCA placebo

SUMMARY:
Phase 3 study to examine whether treatment with ITCA-650 60 mcg/day or 40 mcg/day is superior to placebo when added to current therapy in reducing HbA1c in patients with type 2 diabetes.

ELIGIBILITY:
Inclusion Criteria:

* HbA1c between 7.5% - 10%
* On diet & exercise, metformin (MET), sulfonylurea (SU) or thiazolidinedione (TZD) alone or in combination or combined (SU + TZD) or in combination with Met + SU, Met + TZD, Met + TZD + SU
* BMI between 25 & 45 kg/m2

Exclusion Criteria:

* taking DPP-4 inhibitors, exenatide, liraglutide, alpha glucosidase inhibitors, meglitinides or insulin within last 3 months
* history of pancreatitis

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 460 (Actual)
Dates: Start 2013-03; Primary Completion 2014-08 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Change in HbA1c | 39 weeks
  39-week Treatment Period

CONTACTS AND LOCATIONS:
Locations (105):
- United States (105):
  - Study Site, Birmingham, Alabama
  - Study Site, Gulf Shores, Alabama
  - Study Site, Huntsville, Alabama
  - Study Site, Chandler, Arizona
  - Study Site, Goodyear, Arizona
  - Study Site, Phoenix, Arizona
  - Study Site, Little Rock, Arkansas
  - Study Site, Chula Vista, California
  - Study Site, Fresno, California
  - Intarcia, Hayward, California
  - Study Site, Long Beach, California
  - Study Site, Los Angeles, California
  - Study Site, National City, California
  - Study Site, Port Hueneme, California
  - Study Site, San Jose, California
  - Study Site, San Mateo, California
  - Study Site, Tustin, California
  - Study Site, Valley Village, California
  - Study Site, Walnut Creek, California
  - Study Site, Watsonville, California
  - Study Site, Colorado Springs, Colorado
  - Study Site, Boca Raton, Florida
  - Study Site, Bradenton, Florida
  - Study Site, Celebration, Florida
  - Study Site, Clearwater, Florida
  - Study Site, Coral Gables, Florida
  - Study Site, Daytona Beach, Florida
  - Study Site, Hollywood, Florida
  - Study Site, Jacksonville, Florida
  - Study Site, Miami, Florida
  - Study Site, New Port Richey, Florida
  - Study Site, North Miami Beach, Florida
  - Study Site, Orlando, Florida
  - Study Site, Palm Harbor, Florida
  - Study Site, Pembroke Pines, Florida
  - Study Site, Ponte Vedra, Florida
  - Study Site, Tampa, Florida
  - Study Site, Atlanta, Georgia
  - Study Site, Canton, Georgia
  - Study Site, Idaho Falls, Idaho
  - Study Site, Meridian, Idaho
  - Study Site, Chicago, Illinois
  - Study Site, Evansville, Illinois
  - Study Site, Avon, Indiana
  - Study Site, Evansville, Indiana
  - Study Site, Franklin, Indiana
  - Study Site, Greenfield, Indiana
  - Study Site, Muncie, Indiana
  - Study Site, Valparaiso, Indiana
  - Study Site, Des Moines, Iowa
  - Study Site, Newton, Kansas
  - Study Site, Metaire, Louisiana
  - Study Site, Metairie, Louisiana
  - Study Site, Metarie, Louisiana
  - Study Site, New Orleans, Louisiana
  - Study Site, Baltimore, Maryland
  - Study Site, Brockton, Massachusetts
  - Study Site, Rochester, Michigan
  - Study Site, Ypsilanti, Michigan
  - Study Site, Kansas City, Missouri
  - Study Site, Billings, Montana
  - Study Site, Lincoln, Nebraska
  - Study Site, Las Vegas, Nevada
  - Study Site, Toms River, New Jersey
  - Study Site, Brooklyn, New York
  - Study Site, Endwell, New York
  - Study Site, Staten Island, New York
  - Study Site, Charlotte, North Carolina
  - Study Site, Durham, North Carolina
  - Study Site, Greensboro, North Carolina
  - Study Site, Hickory, North Carolina
  - Study Site, Moorehead City, North Carolina
  - Study Site, Mooresville, North Carolina
  - Study Site, Salisbury, North Carolina
  - Study Site, Wilmington, North Carolina
  - Study Site, Winston-Salem, North Carolina
  - Study Site, Cincinnati, Ohio
  - Study Site, Columbus, Ohio
  - Study Site, Franklin, Ohio
  - Study Site, Toledo, Ohio
  - Study Site, Norman, Oklahoma
  - Study Site, Oklahoma City, Oklahoma
  - Study Site, Bend, Oregon
  - Study Site, Uniontown, Pennsylvania
  - Study Site, Greer, South Carolina
  - Study Site, North Myrtle Beach, South Carolina
  - Study Site, Dakota Dunes, South Dakota
  - Study Site, Knoxville, Tennessee
  - Study Site, Memphis, Tennessee
  - Study Site, Austin, Texas
  - Study Site, Carrolton, Texas
  - Study Site, Corpus Cristi, Texas
  - Study Site, Dallas, Texas
  - Study Site, Fort Worth, Texas
  - Study Site, Houston, Texas
  - Study Site, San Angelo, Texas
  - Study Site, San Antonio, Texas
  - Study Site, Sugar Land, Texas
  - Study Site, Tomball, Texas
  - Study Site, Danville, Virginia
  - Study Site, Norfolk, Virginia
  - Study Site, Richmond, Virginia
  - Study Site, Port Orchard, Washington
  - Study Site, Renton, Washington
  - Study Site, Spokane, Washington

REFERENCES:
- [Derived] Rosenstock J, Buse JB, Azeem R, Prabhakar P, Kjems L, Huang H, Baron MA. Efficacy and Safety of ITCA 650, a Novel Drug-Device GLP-1 Receptor Agonist, in Type 2 Diabetes Uncontrolled With Oral Antidiabetes Drugs: The FREEDOM-1 Trial. Diabetes Care. 2018 Feb;41(2):333-340. doi: 10.2337/dc17-1306. Epub 2017 Dec 14. PMID 29242349